CLINICAL TRIAL: NCT06316076
Title: A Clinical Study for the Safety and Efficacy of CD19-CAR-DNT Cells (RJMty19) in the Treatment of Relapsed or Refractory Autoimmune Diseases
Brief Title: Safety and Efficacy Study of CD19-CAR-DNT Cells in Autoimmune Diseases
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Collaborators: Guangdong Ruishun Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJMty19-AID001
Record Dates: First submitted 2024-03-12; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Systemic Lupus Erythematosus; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Idiopathic Inflammatory Myopathies; Systemic Sclerosis
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Myositis; Scleroderma, Systemic | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19-CAR-DNT cells (Experimental): 8-24 patients are planned to be enrolled in the dose-escalation trial and 12-24 patients in the dose-expansion trial.
  Interventions: Biological: CD19-CAR-DNT cells

INTERVENTIONS:
Biological: CD19-CAR-DNT cells — Lentiviral vector-transduced DNT cells to express anti-CD19 CAR. Prior to cellular infusion, each patient received cyclophosphamide and fludarabine lymphodepleting chemotherapy.
  Other Names: Cyclophosphamide; Fludarabine

SUMMARY:
To evaluate the safety and efficacy of CD19-CAR-DNT cells in subjects with relapsed/refractory autoimmune diseases

DETAILED DESCRIPTION:
This is an open, single-arm, single-dose, dose-escalation and dose-expansion clinical trial designed to evaluate the maximum tolerated dose of CD19-CAR-DNT cells, the safety, the preliminary efficacy and the pharmacokinetic profile of CD19-CAR-DNT cells in patients after infusion. 8-24 patients are planned to be enrolled in the dose-escalation trial and 12-24 patients in the dose-expansion trial. The primary endpoints are DLT, MTD, and the incidence of abnormalities in AE/SAE/AESI/laboratory test.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign an ICF and expect to complete the study procedures for follow-up examinations and treatment;
2. Aged 18 to 75 years (including cut-offs), regardless of gender;
3. Appropriate organ function, and accordance with the following criteria within 7 days prior to lymphodepleting chemotherapy:

   Coagulation function: a) Fibrinogen ≥1.0 g/L; b) Activated partial thromboplastin time ≤1.5 times the upper limit of normal (ULN); c) Prothrombin time (PT) ≤1.5 times ULN;

   Liver function: a) Glutathione aminotransferase (AST) ≤ 3 times the upper limit of normal (ULN); b) Glutamic aminotransferase (ALT) ≤ 3 times ULN; c) Total bilirubin ≤ 1.5 times ULN, unless the subject has documented Gilbert syndrome. Subjects with Gilbert-Meulengracht syndrome with total bilirubin ≤ 1.5 times ULN may be included;

   Renal function: serum creatinine ≤ 1.5 times ULN, or creatinine clearance ≥ 60 mL/min (see Appendix 2 for Cockcroft-Gault formula);

   Complete blood count: a) Hemoglobin ≥ 80 g/L or hemoglobin maintained at that level following transfusion; b) absolute neutrophil count (ANC) ≥ 1.0×10^9/L; c) A platelet count ≥ 30 x 10^9/L or a platelet count maintained at that level following a platelet transfusion;

   Cardiopulmonary function: left ventricular ejection fraction (LVEF) ≥45%;
4. Female patients with of childbearing potential should have a negative pregnancy test during the screening period. Any male and female patients of childbearing potential must agree to use an effective contraception method for at least six months from the time that they sign the informed consent form until the end of the cell infusion. Female patients without childbearing potential (meeting at least 1 of the following criteria) is described below:

   1. Have undergone a hysterectomy or bilateral oophorectomy;
   2. Medically recognized as ovarian failure;
   3. Medically recognized as post-menopausal (at least 12 consecutive months of menopause without pathological or physiological cause);
5. Meets the criteria of relapsed/refractory autoimmune diseases in 2022 EULAR/ACR.

Exclusion Criteria:

1. Individuals with a history of severe drug allergies or allergic constitution;
2. Active infectious diseases: such as tuberculosis, central nervous system infection, hepatitis, enteritis, etc.;
3. The following serious diseases: malignant tumor, end-stage renal failure, alveolar hemorrhage requiring mechanical ventilation, acute mononeuritis multiplex, or CNS involvement;
4. Renal disease: creatinine clearance rate < 60mL/min and serum creatinine > 1.5 times ULN within 1 week before lymphodepleting chemotherapy; Patients required hemodialysis or high-dose glucocorticoid therapy (e.g., prednisone (or equivalent) ≥100mg per day) within 6 months before screening;
5. Cardiovascular disease: unstable angina, cerebrovascular accident or transient ischemic attack, myocardial infarction, New York Heart Association class III or IV cardiac dysfunction, or refractory hypertension within 6 months before screening (refractory hypertension was defined as: on the basis of lifestyle modification, patients were treated with adequate and reasonably tolerable doses of ≥3 antihypertensive drugs (including diuretics) for > 1 month or with ≥4 antihypertensive drugs for effective blood pressure control) and a history of severe arrhythmia requiring drug treatment;
6. Other uncontrollable diseases: clinically unstable or not effectively controlled acute/chronic diseases unrelated to AID (such as acute pneumonia, diabetic ketoacidosis, acute pancreatitis, etc.) that may confound study results or affect investigators' assessment of efficacy/safety;
7. Patients with positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) and peripheral blood hepatitis B virus (HBV) DNA titration assay not within the normal reference range, positive hepatitis C virus (HCV) antibody and peripheral blood HCV RNA, positive for human immunodeficiency virus (HIV), or positive for cytomegalovirus (CMV) DNA, or positive syphilis test;
8. The presence of active or uncontrollable infections requiring systemic treatment (except simple urinary tract infections or upper respiratory tract infections) and currently receiving suppressive therapy for any chronic infection (e.g., tuberculosis, Pneumocystis carinii, cytomegalovirus, herpes simplex virus, herpes zoster, and atypical mycobacteria);
9. Vaccination with live or attenuated live vaccine within 1 month before screening;
10. Persons who have previously received an organ transplant or are preparing to receive an organ transplant;
11. Patients have received CAR-T therapy or other gene-modified cell therapy prior to enrolment;
12. Received rituximab treatment within 6 months prior to screening; Received belimumab and telitacicept within 30 days prior to initial administration of the investigational drug; JAK inhibitor discontinuation time is less than 5 half-lives;
13. Patients with a life expectancy of less than 3 months;
14. Patients have been involved in other clinical studies within 3 months prior to screening;
15. Patients, in the judgement of the investigator and/or clinical criteria, are contraindicated to any study procedure or have other medical conditions that may place them at unacceptable risk.

    -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
DLT | Up to 28 days
  To evaluate the safety, tolerability, and determine the recommended dosage of CD19-CAR-DNT Cell Therapy for Relapsed/Refractory autoimmune disease.
MTD | Up to 28 days
  MTD was the highest dose for DLT in ≤1/6 subjects.
Incidence of abnormalities | Up to 28 days
  Incidence of abnormalities in AE/SAE/AESI/laboratory tests/electrocardiograms/vital signs.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) indicator (Cmax) | Up to 90 days
  The peak concentration of CD19-CAR-DNT cells amplified in the peripheral blood (Cmax, detected by qPCR).
Pharmacokinetics (PK) indicator (AUC) | Up to 90 days
  CD19-CAR-DNT cells blood concentrations will be measured at different time points to evaluate the area under the curve (AUC). (AUC, detected by qPCR)
Pharmacokinetics (PK) indicator (Tmax) | Up to 2 years
  CD19-CAR-DNT cells blood concentrations will be measured at different time points to evaluate the peak plasma time (Tmax). Tmax is defined as the time to reach the highest concentration (Tmax, detected by qPCR).
Pharmacokinetics (PK) indicator (T1/2) | Up to 90 days
  CD19-CAR-DNT cells blood concentrations will be measured at different time points to evaluate the elimination half-life in hours (T1/2). T1/2 is defined as the time point when the concentration of CD19-CAR-DNT reaches half of maximum in a patient's peripheral blood (T1/2, detected by qPCR).
Disease response rate at 6 months | Up to 6 months
  Proportion of subjects with complete or partial remission.
Duration of Response | Up to 2 years
  The time from the first assessment of remission or partial remission of the disease to the first assessment of disease progression or death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rheumatology, Ren Ji Hospital South Campus, School of Medicine, Shanghai JiaoTong University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No